CLINICAL TRIAL: NCT03142100
Title: Assessment of the Contribution of Combined Acoustic Hearing Via a Hearing Aid and Electric Hearing Via a Cochlear Implant in Adult Bimodal Users Following Using a HA With a Dedicated Bimodal Fitting Formula
Brief Title: Combined Acoustic and Electric Hearing (CI/HA) in Adult Bimodal Users Using a HA With a Bimodal Fitting Formula
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Bnai Zion Medical Center (Other Government)
Responsible Party: Principal Investigator, MICAL.LUNTZ, professor, Bnai Zion Medical Center
Other Study IDs: 0097-16
Record Dates: First submitted 2017-02-19; First posted 2017-05-05 (Actual); Last update posted 2017-05-05 (Actual); Status verified 2017-05

CONDITIONS: Hearing Loss
MeSH Terms: conditions — Hearing Loss | interventions — Cochlear Implants; Hearing Aids

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Hebrew speaking participants: Hebrew speaking bilateral-bimodal users will be assessed using cochlear implants and hearing aids
  Interventions: Device: cochlear implants and hearing aids
- Arabic speaking participants: Arabic speaking bilateral-bimodal users will be assessed using cochlear implants and hearing aids
  Interventions: Device: cochlear implants and hearing aids

INTERVENTIONS:
Device: cochlear implants and hearing aids — speech perception tests and bimodal fitting

SUMMARY:
Introduction: Bilateral-bimodal users may benefit from bilateral-binaural and a bimodal effect . The two modes of stimulation complement each other and may overcome the limitation of electric hearing alone. However, alongside the expected benefits of having two hearing systems in bilateral bimodal hearing, there are several inherent mismatches in combing two different stimulation methods, which may negatively impact the processing of the binaural cues.

Aim: To determine whether bimodal listening with a hearing aid programmed using a dedicated bimodal fitting formula, which aligns the frequency response, loudness growth functions, and automatic gain control (AGC) characteristics between the cochlear implant speech processor and the hearing aid brings additional benefit over bimodal listening with the subject's clinical hearing instrument via the use of using a comprehensive battery of speech perception tests aimed at different aspects of binaural hearing as well as the contribution of the unique bimodal complementary effect. A secondary goal is to identify the tests that are best suited to predicting and evaluating bimodal benefit.

Method: The study will include 20 Hebrew and 20 Arabic speakers' adult bilateral-bimodal users that their audiometric thresholds in the non implanted ear will be no worse than 75 dB HL at 250 and 85 dB HL at 500 Hz, who use their hearing aids for at least 75% of their waking hours. The added benefit of the hearing aid programmed using a dedicated bimodal fitting formula will be evaluated using six task-specific tests designed to sensitively assess the bilateral-binaural and bimodal complementary effects using roving speech and noise and different types of background noises (maskers), pitch-related task and subjective questionnaire. Participants will be tested twice in quick succession, at two-weekly intervals, in establishing a baseline score with their clinical HAs. Then participants will be tested again twice in quick succession, at two-weekly intervals following three month experience with the HA fitted with the bimodal fitting formula. All tests will be administered the CI/HA listening condition.

DETAILED DESCRIPTION:
Introduction: Bilateral-bimodal hearing, cochlear implant on one ear and hearing aid on the other ear (CI/HA) may benefit from bilateral-binaural effects as a result of using two hearing systems, and a bimodal effect as a result of using two modes of stimulation, namely acoustic via a HA and electrical via a CI. The two modes of stimulation complement each other and may overcome the limitation of electric hearing alone. However, alongside the expected benefits of having two hearing systems in bilateral bimodal hearing, there are several inherent mismatches in combing two different stimulation methods, which may negatively impact the processing of the binaural cues. These mismatches include mismatch in the incoming speech signal timing; mismatch in pitch balance between two devices, mismatch in the frequency range conferred, and mismatch in the frequency range conveyed to a specific location in the cochlea by the cochlear implant and to a different location in the contra-lateral cochlea by the hearing aid.

Aim: To determine whether bimodal listening with a hearing aid programmed using a dedicated bimodal fitting formula, which aligns the frequency response, loudness growth functions, and automatic gain control (AGC) characteristics between the cochlear implant speech processor and the hearing aid brings additional benefit over bimodal listening with the subject's clinical hearing instrument via the use of using a comprehensive battery of speech perception tests aimed at different aspects of binaural hearing as well as the contribution of the unique bimodal complementary effect. A secondary goal is to identify the tests that are best suited to predicting and evaluating bimodal benefit.

Method: The study will include 20 Hebrew and 20 Arabic speakers' adult bilateral-bimodal users that their audiometric thresholds in the non implanted ear will be no worse than 75 dB HL at 250 and 85 dB HL at 500 Hz, who use their hearing aids for at least 75% of their waking hours. The added benefit of the hearing aid programmed using a dedicated bimodal fitting formula will be evaluated using six task-specific tests designed to sensitively assess the bilateral-binaural and bimodal complementary effects using roving speech and noise and different types of background noises (maskers), pitch-related task and subjective questionnaire. Participants will be tested twice in quick succession, at two-weekly intervals, in establishing a baseline score with their clinical HAs. Then participants will be tested again twice in quick succession, at two-weekly intervals following three month experience with the HA fitted with the bimodal fitting formula. All tests will be administered the CI/HA listening condition.

Data analysis: Speech perception test results and self-rating questionnaire scores will be analyzed by repeated measure analysis of variance. The difference between the two moods of bimodal listening (clinical HA versus HA fitted by the bimodal formula) will be evaluated. Correlation between audiological variables aided and unaided hearing thresholds in the non-implanted ear and the bilateral-bimodal benefit will be examined as well.

ELIGIBILITY:
Inclusion Criteria:

Two groups, ideally each of 20 experienced adult bimodal users will be studied: one Arabic speaking and the other Hebrew speaking.

B. Inclusion criteria:

* Regular adults bimodal users (at least 18 years of age) having continuous use of both CI and hearing instrument for 75% of waking hours.
* Their audiometric thresholds in the non implanted ear will be no worse than 75 dB HL at 250 and 85 dB HL at 500 Hz.
* All participants will have stable CI map and acquired at least twelve month's experience using a CI and HA in combination using the Naida CI sound processor
* Participants will be first language speakers of either Arabic or Hebrew
* Participants will be required to demonstrate highly reliable responses, and will be able to understand recorded speech material in the presence of competing noise, achieving at least 50% correct for sentences when the signal-to-noise-ratio is +20 dB.
* No participant shall have any additional physical or cognitive problem that might interfere with their ability to participate in the study.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study will include 20 Hebrew and 20 Arabic speakers' adult bilateral-bimodal users that their audiometric thresholds in the non implanted ear will be no worse than 75 dB HL at 250 and 85 dB HL at 500 Hz, who use their hearing aids for at least 75% of their waking hours.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2017-06-15 (Estimated); Primary Completion 2019-04-01 (Estimated); Study Completion 2019-06-15 (Estimated)

PRIMARY OUTCOMES:
outcome measure: the speech perception test battery and questionnaire scores will be calculated as follows: [(CI+ HA (old version)] - [ CI+HA (new dedicated prescription)]. | about 2 months
  The added benefit of the hearing aid programmed using a dedicated bimodal fitting formula will be evaluated using six task-specific tests designed to sensitively assess the bilateral-binaural and bimodal complementary effects using roving speech and noise and different types of background noises (maskers), pitch-related task and subjective questionnaire. Participants will be tested twice in quick succession, at two-weekly intervals, in establishing a baseline score with their clinical HAs. Then participants will be tested again twice in quick succession, at two-weekly intervals following three month experience with the HA fitted with the bimodal fitting formula. All tests will be administered in the CI/HA listening condition. Comparison between these test results will estimate the added benefit of the dedicated bimodal formula.

IPD SHARING:
Plan to Share IPD: Undecided